CLINICAL TRIAL: NCT00498004
Title: Randomized, Open Label, 8-Week Study of Quetiapine and Risperidone on Quality of Life in Female With Schizophrenia
Brief Title: Quality of Life (QOL) in Female Patient With Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficult to recruit subject
Sponsor: Inje University (Other)
Responsible Party: Joo Shim, Inje University, Busan Paik Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QOL Study 2007
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-11

CONDITIONS: Schizophrenia
Keywords: Quality of Life; Schizophrenia; Quetiapine; Risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Quetiapine, Risperidone — The dose of quetiapine will be titrated over 4 days to 300mg/day (50mg at day 1, 100mg at day 2, 200mg at day 3 and 300mg at day 4) and thereafter flexible dose will be administered depending on the clinical state. The dose of risperidone will be titrated as following 2mg at day 1 and 4mg at day 4 and thereafter flexible dose will be administered depending on the clinical state. The dosage of drugs should be 400-800mg/day of quetiapine and 4-6mg/day of risperidone between 6 and 8 weeks of trial.

SUMMARY:
The primary objective of this study is to demonstrate clinical and statistical superiority of quetiapine compared to risperidone in Korean version of Heinrich's Quality of Life Scale after 8 weeks trial of drugs.

DETAILED DESCRIPTION:
Prolactin related adverse events are closely related to patient's perception on their illness and quality of life . Poor subjective wellbeing induced by prolactin elevation after antipsychotic drug treatment can complicate the clinical outcomes of treatment.Quetiapine has negligible effects on the elevation of prolactin and does not produce hyperprolactinemia related adverse events such as amenorrhea, galactorrhea that may disturb quality of life in famel patient. In this Randomized, Open Label, 8-week Study, the impact of quetiapine and risperidone on quality of life in female patients with schizophrenia will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Schizophrenia (DSM-IV)
2. Female, Age: between 18-60 years
3. Who either need first time treatment with antipsychotic drug or recently
4. Sign written informed consent

Exclusion Criteria:

1. Taking other psychiatric medications during last 30 days
2. Refractory schizophrenia
3. A current medical illness associated with sexual dysfunction
4. Previous history of no response to quetiapine or risperidone treatment
5. Previous enrolment or randomisation of treatment in the present study.
6. Participation in a clinical study during the last 90 days.
7. Pregnancy
8. Alcohol or substance abuser

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
QOL measured by Korean version of Heinrich's Quality of Life Scale | 8weeks

SECONDARY OUTCOMES:
Korean version of Female Sexual Function Index | 8 weeks
Korean version of Female Sexual Distress Scale | 8 weeks
Hormonal levels (Prolactin, Estradiol, Free Testosterone, FSH, LH | 8 weeks
Psychopathology (Brief Psychiatric Rating Scale) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Cheol Shim, MD,PhD, Principal Investigator — Clinical Trial Center, Paik hospital
Locations (1):
- Busan Paik Hospital, Busan, South Korea

REFERENCES:
- [Background] Jung DU, Conley RR, Kelly DL, Kim DW, Yoon SH, Jang JH, Shin JG, Shim JC. Prevalence of bone mineral density loss in Korean patients with schizophrenia: a cross-sectional study. J Clin Psychiatry. 2006 Sep;67(9):1391-6. doi: 10.4088/jcp.v67n0909. PMID 17017825